CLINICAL TRIAL: NCT00109408
Title: A Randomized, Double-blind Study of Safety and Reduction in Signs and Symptoms During Treatment With Tocilizumab Monotherapy Versus Methotrexate Monotherapy in Patients With Moderate to Severe Active Rheumatoid Arthritis
Brief Title: A Study to Assess the Safety and Efficacy of Tocilizumab in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA17824
Record Dates: First submitted 2005-04-27; First posted 2005-04-28 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]
- 2 (Active Comparator)
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — 7.5-20mg po weekly
  Arms: 2
Drug: tocilizumab [RoActemra/Actemra] — 8mg/kg iv every 4 weeks
  Arms: 1

SUMMARY:
This 2 arm study will assess the safety and efficacy of tocilizumab monotherapy versus methotrexate in patients with active rheumatoid arthritis (RA). Patients will be randomized to receive tocilizumab 8mg/kg iv every 4 weeks plus placebo po weekly, or methotrexate 7.5-20mg po weekly plus placebo iv every 4 weeks. The anticipated time on study treatment is 3-12 months and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients at least 18 years of age with active RA for at least 3 months;
* patients of reproductive potential must be using reliable methods of contraception.

Exclusion Criteria:

* major surgery (including joint surgery) within 8 weeks before entering study or planned major surgery within 6 months after entering study;
* treatment with methotrexate (MTX) within 6 months of entering study;
* patients who have stopped previous MTX treatment due to toxicity or lack of response;
* women who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 673 (Actual)
Dates: Start 2005-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with ACR 20 response | Week 24

SECONDARY OUTCOMES:
Percentage of patients with ACR 20 response | Week 8
Percentage of patients with ACR 50 and ACR 70 responses | Week 24
Mean change in parameters of ACR core set | Week 24
AEs, laboratory parameters, vital signs. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (133):
- United States (66):
  - Montgomery, Alabama
  - Mesa, Arizona
  - Paradise Valley, Arizona
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Huntington Beach, California
  - Long Beach, California
  - Los Angeles, California
  - Palm Springs, California
  - Sacramento, California
  - San Leandro, California
  - Santa Maria, California
  - Jupiter, Florida
  - Palm Habor, Florida
  - Palm Harbor, Florida
  - Port Orange, Florida
  - Tampa, Florida
  - Idaho Falls, Idaho
  - Meridian, Idaho
  - Morton Grove, Illinois
  - Springfield, Illinois
  - Indianapolis, Indiana
  - Cedar Rapids, Iowa
  - Des Moines, Iowa
  - Bowling Green, Kentucky
  - Baton Rouge, Louisiana
  - Slidell, Louisiana
  - Greenbelt, Maryland
  - Pittsfield, Massachusetts
  - Grand Rapids, Michigan
  - Kalamazoo, Michigan
  - Lansing, Michigan
  - Eagan, Minnesota
  - Saint Cloud, Minnesota
  - Flowood, Mississippi
  - Tupelo, Mississippi
  - St Louis, Missouri
  - Dover, New Hampshire
  - Nashua, New Hampshire
  - Haddon Heights, New Jersey
  - New Brunswick, New Jersey
  - Albany, New York
  - Syracuse, New York
  - Fayetteville, North Carolina
  - Canton, Ohio
  - Mayfield, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Willow Grove, Pennsylvania
  - Wyomissing, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Greenville, South Carolina
  - Hickory Grove, South Carolina
  - Hixson, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Austin, Texas
  - Mesquite, Texas
  - Chesapeake, Virginia
  - Mountlake Terrace, Washington
  - Olympia, Washington
  - Spokane, Washington
  - Yakima, Washington
- Argentina (3):
  - Buenos Aires
  - Rosario
  - San Juan Bautista
- Australia (6):
  - Adelaide
  - Hobart
  - Shenton Park
  - Sydney
  - Woodville
  - Woolloongabba
- Canada (8):
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Burlington, Ontario
  - Hamilton, Ontario
  - Kitchener, Ontario
  - Mississauga, Ontario
  - Ottawa, Ontario
- China (3):
  - Guangzhou
  - Hefei Anhui
  - Jinan
- Denmark (3):
  - Copenhagen
  - Hillerød
  - Hvidovre
- France (4):
  - Brest
  - Lyon
  - Paris
  - Rouen
- Israel (6):
  - Ashkelon
  - Beersheba
  - Haifa
  - Kfar Saba
  - Ramat Gan
  - Rishon LeZiyyon
- Italy (5):
  - Genova
  - Milan
  - Pavia
  - Reggio Emilia
  - Siena
- Lithuania (5):
  - Kaunas
  - Klaipėda
  - Panevezys
  - Šiauliai
  - Vilnius
- Mexico (2):
  - Guadalajara
  - Mexico City
- Norway (2):
  - Levanger
  - Lillehammer
- Lima, Peru
- Portugal (2):
  - Almada
  - Lisbon
- Serbia (2):
  - Belgrade
  - Niška Banja
- Slovenia (2):
  - Ljubljana
  - Maribor
- South Africa (4):
  - Cape Town
  - Diepkloof
  - Pinelands
  - Radiokop
- Spain (9):
  - Alcorcón
  - Barcelona
  - Córdoba
  - Guadalajara
  - Lugo
  - Salamanca
  - San Cristóbal de La Laguna
  - Santiago de Compostela
  - Valencia

REFERENCES:
- [Derived] Drobinski PJ, Bay-Jensen AC, Karsdal MA, Sardar S, Siebuhr AS. Connective tissue remodelling is differently modulated by tocilizumab versus methotrexate monotherapy in patients with early rheumatoid arthritis: the AMBITION study. Arthritis Res Ther. 2021 Jan 7;23(1):13. doi: 10.1186/s13075-020-02378-7. PMID 33413588
- [Derived] Strand V, Michalska M, Birchwood C, Pei J, Tuckwell K, Finch R, Gabay C, Kavanaugh A, Jones G. Impact of tocilizumab monotherapy on patient-reported outcomes in patients with rheumatoid arthritis from two randomised controlled trials. RMD Open. 2017 Sep 14;3(2):e000496. doi: 10.1136/rmdopen-2017-000496. eCollection 2017. PMID 28955499
- [Derived] Jones G, Wallace T, McIntosh MJ, Brockwell L, Gomez-Reino JJ, Sebba A. Five-year Efficacy and Safety of Tocilizumab Monotherapy in Patients with Rheumatoid Arthritis Who Were Methotrexate- and Biologic-naive or Free of Methotrexate for 6 Months: the AMBITION Study. J Rheumatol. 2017 Feb;44(2):142-146. doi: 10.3899/jrheum.160287. Epub 2016 Dec 1. PMID 27909081
- [Derived] Wang J, Bansal AT, Martin M, Germer S, Benayed R, Essioux L, Lee JS, Begovich A, Hemmings A, Kenwright A, Taylor KE, Upmanyu R, Cutler P, Harari O, Marchini J, Criswell LA, Platt A. Genome-wide association analysis implicates the involvement of eight loci with response to tocilizumab for the treatment of rheumatoid arthritis. Pharmacogenomics J. 2013 Jun;13(3):235-41. doi: 10.1038/tpj.2012.8. Epub 2012 Apr 10. PMID 22491018
- [Derived] Jones G, Sebba A, Gu J, Lowenstein MB, Calvo A, Gomez-Reino JJ, Siri DA, Tomsic M, Alecock E, Woodworth T, Genovese MC. Comparison of tocilizumab monotherapy versus methotrexate monotherapy in patients with moderate to severe rheumatoid arthritis: the AMBITION study. Ann Rheum Dis. 2010 Jan;69(1):88-96. doi: 10.1136/ard.2008.105197. PMID 19297346